CLINICAL TRIAL: NCT04091880
Title: A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Safety and Immunogenicity of Simultaneously Administration of EV71 Vaccine and Influenza Vaccine (Split Virion),Inactivated
Brief Title: Evaluation of the Safety and Immunogenicity of Simultaneously Administration of EV71 Vaccine and Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Henan Center for Disease Control and Prevention (Other Government); Guizhou Center for Disease Control and Prevention (Other); Wuhan Institute of Biological Products Co., Ltd (Industry); Changchun Institute of Biological Products Co., Ltd. (Industry); Peking University (Other); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EV71-Flu-Combine-01
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Enterovirus Infections; Influenza
Keywords: EV71 vaccine; influenza vaccine; simultaneously administration
MeSH Terms: conditions — Enterovirus Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): 378 subjects from the experimental group will be simultaneously administrated with one dose of EV71 vaccine (0.5 ml) and one dose of influenza vaccine (0.25 ml). One month later, they are going to receive a second dose of EV71 vaccine and influenza vaccine, simultaneously.
  Interventions: Biological: EV71 vaccine and influenza vaccine
- control group A (Active Comparator): 378 subjects from the control group A will be only administrated with two doses of EV71 vaccine (0.5 ml) (1 month apart).
  Interventions: Biological: EV71 vaccine
- control group B (Active Comparator): 378 subjects from the control group B will be only administrated with two doses of influenza vaccine (0.25 ml) (1 month apart).
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: EV71 vaccine and influenza vaccine — simultaneously administrated with EV71 vaccine and influenza vaccine
  Arms: experimental group
Biological: EV71 vaccine — administrated with EV71 vaccine only
  Arms: control group A
Biological: influenza vaccine — administrated with influenza vaccine only
  Arms: control group B

SUMMARY:
Subjects will be recruited and divided into 3 groups:

1. Experimental Group (378 subjects): combined immunization of EV71 vaccine and influenza vaccine;
2. Control Group A (378 subjects): EV71 vaccine only;
3. Control Group B (378 subjects): influenza vaccine only;

All blood samples will be collected before and one month after vaccinatioin. The immunogenicity and safety of both experimental and control groups will be compared and the data be analyzed.

DETAILED DESCRIPTION:
To further evaluate the feasibility of simultaneously administration of EV71 vaccine and flu vaccine, we design this clinical trial to test its immunogenicity and safety. 1134 subjects aged from 6 to 11 months old are divided into one experimental group and two control groups (control group A and B).

378 subjects from the experimental group will be simultaneously administrated with one dose of EV71 vaccine (0.5 ml) and one dose of influenza vaccine (0.25 ml). One month later, they are going to receive a second dose of EV71 vaccine and influenza vaccine, simultaneously. Blood samples are collected before the first vaccination, and one month following the second vaccination.

378 subjects from the control group A will be only administrated with two doses of EV71 vaccine (0.5 ml) (1 month apart). Blood samples are collected before the first vaccination, and one month following the second vaccination.

378 subjects from the control group B will be only administrated with two doses of influenza vaccine (0.25 ml) (1 month apart). Blood samples are collected before the first vaccination, and one month following the second vaccination.

To evaluate the immunogenicity, we will detect and compare the neutralization antibody levels, the seroprotection rates, and antibody geometric mean concentrations. The safety of all groups will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged from 6-11 months old at the date of recruitment;
* with informed consent signed by parent(s) or guardians;
* parent(s) or guardians are able to attend all planned clinical appointments and comply with all study instructions;
* subjects not receive any vaccination within 14 days at the date of recruitment;
* subjects have not been vaccinated with EV71 vaccine, seasonal flu vaccine;
* subjects with no medical history of EV71 infection;
* axillary temperature ≤37.0℃

Exclusion Criteria:

* subject who has a medical history with Hypersensitiveness, eclampsia, epilepsy, cerebropathia and neurological illness;
* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* subjects with immunodeficency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(Taking orally injecting of steroid hormone);
* administration of immunoglobulins within 30 days prior to this study;
* acute febrile disease(temperature ≥ 37.0°C) or infectious disease;
* have a clearly diagnosed history of thrombocytopenia or other coagulopathy,
* may cause contraindications for subcutaneous injection;
* any serious chronic illness, acute infectious diseases, or respiratory diseases;
* severe cardiovascular disease, liver and kidney diseases or diabetes mellitus with complications;
* any kind of infectious, purulent, or allergic skin diseases;
* any other factor that makes the investigator determines the subject is unsuitable for this study.

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1134 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate I | Baseline (before vaccination) and 1 month after the last dose
  the rate of positive seroconversion against EV71
Seroconversion rate II | Baseline (before vaccination ) and 1 month after the last dose
  the rate of positive seroconversion against Influenza A (H3N2, H1N1) and B Type viruses
Geometric mean titer (GMT) I | Baseline (before vaccination) and 1 month after the last dose
  Measure neutralizing antibody titers against EV71
Geometric mean titer (GMT) II | Baseline (before vaccination) and 1 month after the last dose
  Measure neutralizing antibody titers against Influenza A (H3N2, H1N1) and B Type viruses

SECONDARY OUTCOMES:
adverse events following vaccination | 6 months
  analyse the numbers and rates of participants who experience adverse events following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Xiao Y, Ye Y, Jiang F, He H, Luo L, Chen H, Shi L, Mu Q, Chen W, Guo X, Zhang M, Li J, Guan Q, Chen Z, Yang X. Immunogenicity and safety of an inactivated enterovirus 71 vaccine coadministered with trivalent split-virion inactivated influenza vaccine: A phase 4, multicenter, randomized, controlled trial in China. Front Immunol. 2022 Dec 8;13:1080408. doi: 10.3389/fimmu.2022.1080408. eCollection 2022. PMID 36569946